CLINICAL TRIAL: NCT07361653
Title: A Prospective, Global, Multicenter, Randomized, Double Blind, Sham Controlled Study to EValuate the Safety and effectIVEness of the Ryme Medical Targeted Lung Denervation (TLD) Catheter in Patients With Moderate and Severe Symptomatic Chronic Obstructive Pulmonary Disease (COPD) - The REVIVE Pivotal Study
Brief Title: The REVIVE Pivotal Study
Acronym: REVIVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ryme Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-01
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); COPD Exacerbations; COPD Patients; COPD Acute Exacerbation; COPD; Lung Disease Airways; Lung Disease, Chronic Obstructive
Keywords: COPD; Targeted Lung Denervation; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Ryme Targeted Lung Denervation (TLD) Procedure (Experimental): Ryme TLD Procedure
  Interventions: Device: Ryme TLD
- Sham Control Procedure (Sham Comparator): Sham Control Procedure
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: Ryme TLD — Ryme TLD Procedure
  Arms: Ryme Targeted Lung Denervation (TLD) Procedure
Device: Sham Control — Sham Control Procedure
  Arms: Sham Control Procedure

SUMMARY:
The goal of this study is to test whether a new treatment called the Ryme Medical Targeted Lung Denervation (TLD) Catheter is safe and effective for people with moderate to severe chronic obstructive pulmonary disease (COPD).

The main questions it aims to answer are:

1. Does the TLD Catheter improve symptoms in people with COPD?
2. Is the TLD Catheter safe ?

Researchers will compare the group receiving the TLD treatment to the group receiving a sham procedure to see if the treatment improves quality of life.

Participants will:

1. Be randomly assigned to receive either the TLD treatment or a sham procedure.
2. Undergo the assigned procedure in a hospital setting.
3. Attend follow-up visits for health checks and breathing tests.

DETAILED DESCRIPTION:
This study is a prospective, global, multicenter, randomized, double blind, sham controlled study to evaluate the safety and effectiveness of the Ryme Medical Targeted Lung Denervation (TLD) Catheter compared to sham in patients with moderate and severe symptomatic chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic chronic obstructive pulmonary disease
* History of COPD exacerbation(s)
* Stable medical therapy
* Candidate for bronchoscopy

Exclusion Criteria:

* Prior lung intervention with device in place
* Using tobacco products, e-cigarettes, vape or other inhaled non-pharmacological substance
* Clinically significant serious or unstable medical conditions (e.g., heart disease requiring treatment, uncontrolled diabetes)
* Pregnant, nursing, or intent to become pregnant during study duration

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) | 12 months
  Change from baseline

SECONDARY OUTCOMES:
St. George Respiratory Questionnaire (SGRQ) Total Score | 12 months
  Change from baseline
Six Minute Walk Test (6MWT) | 12 months
  Change from baseline
COPD exacerbations | 12 months
  Rate of severe post-treatment COPD exacerbations

IPD SHARING:
Plan to Share IPD: No